CLINICAL TRIAL: NCT06133712
Title: A Comparative Study Between Dexmedetomidine, Ozone and Dexamethasone Local Injection in Carpal Tunnel Syndrome for Long- Term Pain Relief
Brief Title: Dexmedetomidine, Ozone and Dexamethasone Local Injection in Carpal Tunnel Syndrome for Pain Relief
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mahmoud T Elgebaly,MD, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36226/12/22
Record Dates: First submitted 2023-11-02; First posted 2023-11-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel; Dexmedetomidine; Ozone; Dexamethasone
MeSH Terms: conditions — Median Neuropathy | interventions — Dexmedetomidine; Ozone; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Active Comparator): Patients will receive injection of 1 microgram/kg dexmedetomidine average (70-100-microgram) (0.7-1ml) plus 4ml lidocaine injection nearby median nerve
  Interventions: Drug: Dexmedetomidine
- Ozone (Active Comparator): Participants will receive a single local injection of 4 ml ozone (10 micrograms/ml) plus to 1 ml lidocaine (1%) using a 25 G needle.
  Interventions: Drug: Ozone
- Dexamethasone (Active Comparator): Patients will receive a single local injection of 5 mL (3 mL lidocaine (1%) and 2 mL [8 mg] dexamethasone) via the same technique.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive injection of 1 microgram/kg dexmedetomidine average (70-100-microgram) (0.7-1ml) plus 4ml lidocaine injection nearby median nerve.
  Other Names: Precedex®
  Arms: Dexmedetomidine
Drug: Ozone — Participants will receive a single local injection of 4 ml ozone (10 micrograms/ml) plus to 1 ml lidocaine (1%) using a 25 G needle.
  Other Names: PubChem CID 24823
  Arms: Ozone
Drug: Dexamethasone — Patients will receive a single local injection of 5 mL (3 mL lidocaine (1%) and 2 mL [8 mg] dexamethasone) via the same technique.
  Other Names: Decadron
  Arms: Dexamethasone

SUMMARY:
The aim of the present study is to compare the analgesic efficacy of Dexmedetomidine, Ozone and Dexamethasone regional injection in carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a collection of symptoms and signs associated with median neuropathy at the carpal tunnel. Most CTS is related to idiopathic compression of the median nerve as it travels through the wrist at the carpal tunnel.

Corticosteroid injection is an extensively used and accepted treatment in mild to moderate CTS according to the guidelines of the American Academy of Orthopedic Surgeons as corticosteroids reduce the inflammation and edema associated with CTS. However, there is no guideline as to which corticosteroid has to be used as the standard treatment in CTS.

Triamcinolone acetonide, a commonly used steroid for this indication, is a particulate steroid, which can cause permanent nerve injury if accidentally injected into the nerve.

Local ozone injection as a therapeutic option in some musculoskeletal conditions; ozone (O3) gas is a molecule consisting of three oxygen atoms in a dynamically unstable structure. Ozone therapy has been utilized and studied for more than a century.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 60 years.
* Both sexes.
* Patients with ultrasonographic evidence of mild-to-moderate carpal tunnel syndrome (CTS).
* Inclusion criteria will include numbness and pain in the median nerve (MN) distribution persisting for minimum of 3 months , nerve conduction studies (NCS) consistent with carpal tunnel syndrome (CTS) as per the American Association of Neuromuscular and Electro diagnostic Medicine (AANEM) guidelines, and an median nerve (MN) cross-sectional area (CSA)at the wrist >12 mm2 suggesting mild-to-moderate CTS forms.

Exclusion Criteria:

* Patient refusal.
* Patients with severe symptoms and signs of CTS as identified per the American Association of Neuromuscular and Electro diagnostic Medicine (AANEM) guidelines,[14] as this is an indication for surgery,
* Patients who show improvement on medical treatment,
* Previous surgical or injectional CTS treatment,
* Pregnancy ,co existence of brachial plexopathy, or thoracic outlet syndrome, polyneuropathy, radiculopathy and peripheral nerve lesion in upper limb.
* Severe cardiovascular disease
* Morbid obese patients (body mass index (BMI) of >35 kg/m2)
* Infection at site of injection.
* Bleeding diathesis.
* History of thyroid deficiency, uncontrolled diabetes mellitus , rheumatoid arthritis and history of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* History of Ozone or Dexmedetomidine allergy.
* End stage renal and hepatic disease.
* History of inflammatory joint , connective tissue disorders, , burns, any local tissue contractures and history of wrist trauma.
* Patients who will not consent to completing The visual analogue scale (VAS) for pain or nerve conduction study before and after injection.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The analgesic efficacy and functional status improvement of Dexmedetomidine, Ozone and Dexamethasone regional injection in carpal tunnel syndrome | Each patient will be assessed at the baseline (before injection) , at 1week, 4weeks, 12weeks, and 24weeks intervals after injection date
  The analgesic efficacy and functional status improvement of Dexmedetomidine, Ozone and Dexamethasone regional injection in carpal tunnel syndrome via assessment of Visual Analogue Scale (VAS) before and after injection.
  VAS used as an effective tool to detect intensity of pain will be recorded (0 to10) "0" represents no pain ,"10" worst pain, "1-3" mild pain,"4-6 " moderate pain and" 7-10 " severe pain.
  Each patient will be assessed at the baseline (before injection) , at 1week, 4weeks, 12weeks, and 24 weeks intervals after injection.

SECONDARY OUTCOMES:
Median motor nerve conduction study(NCS) evaluation | Each patient will be assessed at the baseline (before injection) , at 1week, 4weeks, 12weeks, and 24weeks intervals after injection date
  Each patient will be assessed regarding electrophysiological changes sensory nerve conduction velocity in millimeter/seconds and distal motor latency in milliseconds at the baseline (before injection), at 1week, 4weeks, 12 weeks and 24 weeks intervals after injection.
Sensory nerve conduction study(NCS) evaluation | Each patient will be assessed at the baseline (before injection) , at 1week, 4weeks, 12weeks, and 24weeks intervals after injection date
  Each patient will be assessed regarding electrophysiological changes sensory nerve conduction velocity in millimeter/seconds and distal motor latency in milliseconds at the baseline (before injection), at 1week, 4weeks, 12weeks, and 24 weeks intervals after injection.
Analgesic requirement | First 48 hours post injection .
  Analgesic requirement ( dose and frequency of oral acetaminophen intake in first 48 hours) for post injection .

CONTACTS AND LOCATIONS:
Overall Officials: MAHMOUD ELGEBALY, MD, Principal Investigator — Tanta faculty of medicine
Locations (1):
- Faculty of Medicine, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

DOCUMENTS (1):
  • Study Protocol (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT06133712/Prot_000.pdf